CLINICAL TRIAL: NCT00076960
Title: Compassionate Use of Stannsoporfin as an Adjuvant to Phototherapy to Reduce the Need for Exchange Transfusions
Brief Title: Compassionate Use of Stanate (TM) [Stannsoporfin]
Status: No longer available | Type: Expanded Access
Sponsor: InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Other Study IDs: 99A; NCT01183988 (obsolete NCT alias)
Record Dates: First submitted 2004-02-06; First posted 2004-02-10 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2016-01

CONDITIONS: Neonatal Jaundice; Hyperbilirubinemia
Keywords: hyperbilirubinemia; jaundice; tin-mesoporphyrin; stannsoporfin; exchange transfusion; neonatal hyperbilirubinemia
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia; Jaundice; Hyperbilirubinemia, Neonatal | interventions — tin mesoporphyrin

INTERVENTIONS:
Drug: Stanate (TM) [stannsoporfin, tin-mesoporphyrin] — Treatment with 4.5 mg/kg

SUMMARY:
The purpose of this protocol is to make Stanate (TM) [stannsoporfin, tin-mesoporphyrin] available to infants who meet the following criteria:

1. the infant has a very high level of bilirubin without an adequate clinical response to phototherapy;
2. the infant requires an exchange transfusion; and
3. the family refuses to allow the administration of blood products, particularly on religious grounds, such as within the Jehovah's Witness community.

ELIGIBILITY:
* Term or near term neonate
* Elevated serum bilirubin
* Failing phototherapy
* Requires exchange transfusion
* Family refuses exchange transfusion on religious grounds

Ages: 12 Hours to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

REFERENCES:
- [Background] Kappas A, Drummond GS, Munson DP, Marshall JR. Sn-Mesoporphyrin interdiction of severe hyperbilirubinemia in Jehovah's Witness newborns as an alternative to exchange transfusion. Pediatrics. 2001 Dec;108(6):1374-7. doi: 10.1542/peds.108.6.1374. PMID 11731664